CLINICAL TRIAL: NCT04603170
Title: University of Bojnord
Brief Title: Relationships of Executive Functions, Severity of Psychiatric Symptoms With Response to Therapy
Status: Completed | Type: Observational
Sponsor: Malahat Amani (Other)
Responsible Party: Sponsor-Investigator, Malahat Amani, Malahat Amani, University of Bojnord
Organization: University of Bojnord (Other)
Other Study IDs: 13180899
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Patient Acceptance of Health Care
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: DRUG — taking drug medication prescribed by psychiatrists for at least one month

SUMMARY:
This study was conducted to investigate the moderating role of executive functions in the relationship between the severity of psychiatric symptoms and response to therapy. The statistical population of this study was all outpatients with anxiety disorders and depression who referred to psychiatric clinics.

DETAILED DESCRIPTION:
This study was conducted to investigate the moderating role of executive functions in the relationship between the severity of psychiatric symptoms and response to drug therapy in depressed and anxious patients. The statistical population of this study was all outpatients with anxiety disorders and depression who referred to psychiatric clinics. 164 participants completed Outcome Questionnaire, Brief Symptom Inventory, and Behavior Rating Inventory of Executive Function (BRIEF).

ELIGIBILITY:
Inclusion Criteria:

receiving a diagnosis of anxiety and depression disorders, age over 18 years, and taking drug medication prescribed by psychiatrists for at least one month.-

Exclusion Criteria:

* having psychotic disorders, age under 18 years and absence from treatment.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The statistical population included all adult outpatients with anxiety and depression disorders who referred to psychiatric offices in Bojnord city Sample was selected among the clients of psychiatric offices who received the diagnosis of anxiety and depression disorders and volunteer to participate in the study were sample (n=164)
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Outcome questionnaire | ONE WEEK
  This questionnaire was designed to assess response to treatment. This questionnaire has the dimension of mental distress or signs of distress, interpersonal relationships, and social role. This 45-item questionnaire is answered on a 5-point Likert scale ranging 0 to 4 (not at all to extremely).Scores range from 0 to180. higher scores mean a worse outcome.
Brief Symptom Inventory | ONE WEEK
  This inventory measures the symptoms of psycho-somatization, obsessive-compulsive, interpersonal sensitivity, paranoid thoughts, depression, psychosis, general anxiety, hostility and anxiety. It was answered to questions based on the 5-point Likert scale ranging from 0 to 4 (not at all to perfectly). This questionnaire is 53 items. Scores range from 0 to 212.range of score are higher scores mean a worse outcome and mental health problems.
Behavior Rating Inventory of Executive Function | ONE WEEK
  This questionnaire is used to measure the executive functions of adults aged 18 to 90 from their daily performance in the natural environment. It has 75 items that measure factors including response inhibition, shifting, emotional control, self-monitoring, initiation, working memory, planning, material organization, and task monitoring. It was answered to questions based on the 3-point Likert scale ranging from 0 to 2 (not at all to extremely). the scores range 0 to 150. High score is indicator of weak executive functions.

CONTACTS AND LOCATIONS:
Overall Officials: Malahat amani, ph.d, Principal Investigator — University of Bojnord
Locations (1):
- Malahat Amani, Bojnourd, North Khorsan, Iran

IPD SHARING:
Plan to Share IPD: No